CLINICAL TRIAL: NCT02248259
Title: Open-label, Randomised, Two-way Crossover Study to Assess the Effect of Once Daily Itraconazole on the Pharmacokinetics of BI 409306 After a Single Oral Dose in Healthy Male Volunteers Genotyped as Poor and Extensive Metabolizers of CYP2C19
Brief Title: Drug Drug Interaction Trial With Strong CYP3A4 Inhibitor (Itraconazole) in CYP2C19 Extensive Metabolizers and Poor Metabolizers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1289.23
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306; Itraconazole

ARMS (4):
- Extensive Metabolisers: Ref / Test (Experimental): Participants who were extensive metabolisers received two treatments in a randomised order, the treatments were:
  * Reference (ref) treatment (1 single tablet of 25 mg BI 409306 taken orally on day 1).
  * Test treatment (2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1.
  Interventions: Drug: BI 409306; Drug: Itraconazole
- Poor Metabolisers: Ref / Test (Experimental): Participants who were poor metabolisers received two treatments in a randomised order, the treatments were:
  * Reference (ref) treatment (1 single tablet of 25 mg BI 409306 taken orally on day 1).
  * Test treatment (2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1.
  Interventions: Drug: BI 409306; Drug: Itraconazole
- Extensive Metabolisers: Test / Ref (Experimental): Participants who were extensive metabolisers received two treatments in a randomised order, the treatments were:
  * Test treatment (2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1.
  * Reference (ref) treatment (1 single tablet of 25 mg BI 409306 taken orally on day 1).
  Interventions: Drug: BI 409306; Drug: Itraconazole
- Poor Metabolisers: Test / Ref (Experimental): Participants who were poor metabolisers received two treatments in a randomised order, the treatments were:
  * Test treatment (2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1.
  * Reference (ref) treatment (1 single tablet of 25 mg BI 409306 taken orally on day 1).
  Interventions: Drug: BI 409306; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 409306 — Oral single dose of BI 409306
Drug: Itraconazole — Oral dose, twice daily on Day -3, once daily on Day -2 to Day 2 of Itraconazole

SUMMARY:
The objective of the current study is to evaluate the effect of once daily itraconazole on the pharmacokinetics of BI 409306 in poor (PM) and extensive metabolisers (EM) of CYP2C19.

ELIGIBILITY:
Inclusion criteria:

- Healthy CYP2C19 genotyped male volunteers according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR, respiratory rate, body temperature), 12-lead ECG, ophthalmologic exam, clinical laboratory tests

* Korean ethnicity according to the following criteria: be a current Korean passport or national identification card holder, and have parents and grandparents who were all born in Korea
* Age 20 or older than 20 and 45 or younger than 45 years
* BMI (Body Mass Index) 18.5 or more than 18.5 and BMI 25 or less than 25 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

* Any finding of the medical examination (including BP, PR, respiratory rate, body temperature and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy, hernia surgery)
* Diseases of the central nervous system (including but not limited to any kind of seizures, migraine, stroke or psychiatric disorders) within the past 6 month
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (longer than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or more than 3 cigars or more than 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 20 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval more than 450 ms)
* A history of additional risk factors for Torsade des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Abnormality on color vision test or any other finding on ophthalmologic exam that is clinically deemed to potentially interfere with the safety assessment of this trial
* Subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two month after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.23.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, open-label, 2-way crossover trial.
  The two treatment periods were separated by a washout period of at least 3 weeks.
Period: Treatment Period 1
Arm/Group | Extensive Metabolisers: Ref / Test | Poor Metabolisers: Ref / Test | Extensive Metabolisers: Test / Ref | Poor Metabolisers: Test / Ref
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Extensive Metabolisers: Ref / Test | Poor Metabolisers: Ref / Test | Extensive Metabolisers: Test / Ref | Poor Metabolisers: Test / Ref
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who received at least one dose of trial medication.
Groups:
- Extensive Metabolisers: Participants who were extensive metabolisers received two treatments in a randomised order, the treatments were:
  * Reference (ref) treatment (1 single tablet of 25 mg BI 409306 taken orally on day 1).
  * Test treatment (2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1.
- Poor Metabolisers: Participants who were poor metabolisers received two treatments in a randomised order, the treatments were:
  * Reference (ref) treatment (1 single tablet of 25 mg BI 409306 taken orally on day 1).
  * Test treatment (2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1.
- Total: Total of all reporting groups
Arm/Group | Extensive Metabolisers | Poor Metabolisers | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (8.36) | 29.7 (6.53) | 31.0 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: AUC0-infinity of BI 409306 and Its Metabolites
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) of BI 409306 and its metabolites CD 13896 and CD 14084
Time Frame: 1 hour (h) before drug administration and 10minutes (min), 20min, 30min, 45min, 1h, 1h 30min, 2h, 3h, 4h, 7h, 10h, 12h, 14h, 24h, 48h and 72h (only for test treatment) after drug administration
Population: Pharmacokinetic set (PKS) which included all treated subjects who provided at least one evaluable primary or secondary endpoint in any of the study periods without important protocol violations with respect to the statistical evaluation of relative bioavailability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)*hour (h) /Liter (L)
Groups:
- Extensive Metabolisers: Ref. Treatment: Participants who were extensive metabolisers received 1 single tablet of 25 mg BI 409306 taken orally on day 1 (reference treatment)
- Extensive Metabolisers: Test Treatment: Participants who were extensive metabolisers received 2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1 (test treatment)
- Poor Metabolisers: Ref. Treatment: Participants who were poor metabolisers received 1 single tablet of 25 mg BI 409306 taken orally on day 1 (reference treatment)
- Poor Metabolisers: Test Treatment: Participants who were poor metabolisers received 2 capsules of 100 mg itraconazole taken orally twice daily on day -3 (loading dose) and once daily on day -2 to day 2, plus 1 tablet of 25 mg BI 409306 taken orally as a single dose 1 hour after the itraconazole administration on day 1 (test treatment)
Arm/Group | Extensive Metabolisers: Ref. Treatment | Extensive Metabolisers: Test Treatment | Poor Metabolisers: Ref. Treatment | Poor Metabolisers: Test Treatment
Number analyzed (Participants) | 12 | 12 | 12 | 12
nanomole (nmol)*hour (h) /Liter (L)
  BI 409306 | 547 (71.6) | 621 (68.8) | 1560 (45.5) | 1370 (39.4)
  CD 13896 | 389 (26.4) | 347 (19.2) | 178 (20.0) | 165 (14.3)
  CD 14084 | 2120 (10.9) | 2110 (12.6) | 1810 (15.7) | 1890 (14.2)
Statistical Analysis 1: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for BI 409306; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 113.60, 90% CI 2-sided [100.522 to 128.376], Standard Error of Mean 1.070 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 2: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for BI 409306; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 87.98, 90% CI 2-sided [77.839 to 99.452], Standard Error of Mean 1.070 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment
Statistical Analysis 3: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for CD 13896; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 89.21, 90% CI 2-sided [84.636 to 94.021], Standard Error of Mean 1.029 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 4: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis of CD 13896; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 92.89, 90% CI 2-sided [88.592 to 97.396], Standard Error of Mean 1.026 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment
Statistical Analysis 5: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for CD 14084; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 99.61, 90% CI 2-sided [95.796 to 103.584], Standard Error of Mean 1.022 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 6: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for CD 14084; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 104.37, 90% CI 2-sided [98.783 to 110.278], Standard Error of Mean 1.031 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment

2. Primary Outcome: Cmax of BI 409306 and Its Metabolites
Description: Maximum measured concentration of the analyte in plasma (Cmax) of BI 409306 and its metabolites CD 13896 and CD 14084
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Extensive Metabolisers: Ref. Treatment | Extensive Metabolisers: Test Treatment | Poor Metabolisers: Ref. Treatment | Poor Metabolisers: Test Treatment
Number analyzed (Participants) | 12 | 12 | 12 | 12
nmol/L
  BI 409306 | 264 (67.8) | 246 (60.2) | 564 (50.5) | 432 (35.4)
  CD 13896 | 139 (41.6) | 110 (35.5) | 44.9 (33.3) | 42.8 (16.2)
  CD 14084 | 714 (21.5) | 620 (19.1) | 470 (35.8) | 505 (20.3)
Statistical Analysis 1: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for BI 409306; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 93.26, 90% CI 2-sided [80.377 to 108.217], Standard Error of Mean 1.086 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 2: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for BI 409306; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 76.65, 90% CI 2-sided [60.482 to 97.141], Standard Error of Mean 1.140 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment
Statistical Analysis 3: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for CD 13896; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 78.71, 90% CI 2-sided [67.304 to 92.052], Standard Error of Mean 1.090 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 4: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for CD 13896; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 95.29, 90% CI 2-sided [81.092 to 111.964], Standard Error of Mean 1.093 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment
Statistical Analysis 5: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for CD 14084; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 86.79, 90% CI 2-sided [80.731 to 93.309], Standard Error of Mean 1.041 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 6: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for CD 14084; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 107.45, 90% CI 2-sided [91.764 to 125.812], Standard Error of Mean 1.091 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment

3. Secondary Outcome: AUC0-tz of BI 409306 and Its Metabolites
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable plasma concentration (AUC0-tz) of BI 409306 and its metabolites CD 13896 and CD 14084
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Extensive Metabolisers: Ref. Treatment | Extensive Metabolisers: Test Treatment | Poor Metabolisers: Ref. Treatment | Poor Metabolisers: Test Treatment
Number analyzed (Participants) | 12 | 12 | 12 | 12
nmol*h/L
  BI 409306 | 546 (71.6) | 620 (68.8) | 1560 (45.5) | 1370 (39.4)
  CD 13896 | 388 (26.7) | 345 (19.4) | 176 (20.0) | 163 (14.3)
  CD 14084 | 2120 (11.0) | 2110 (12.6) | 1810 (15.7) | 1890 (14.2)
Statistical Analysis 1: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for BI 409306; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 113.61, 90% CI 2-sided [100.505 to 128.427], Standard Error of Mean 1.070 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 2: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for BI 409306; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 87.91, 90% CI 2-sided [77.763 to 99.370], Standard Error of Mean 1.070 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment
Statistical Analysis 3: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for CD 13896; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 89.05, 90% CI 2-sided [84.478 to 93.859], Standard Error of Mean 1.029 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 4: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for CD 13896; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 92.48, 90% CI 2-sided [88.278 to 96.889], Standard Error of Mean 1.026 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment
Statistical Analysis 5: Comparison: Extensive Metabolisers: Ref. Treatment vs Extensive Metabolisers: Test Treatment; Analysis for CD 14084; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 99.61, 90% CI 2-sided [95.791 to 103.583], Standard Error of Mean 1.022 — Ratio calculated as extensive metabolisers test treatment divided by extensive metabolisers: ref. treatment
Statistical Analysis 6: Comparison: Poor Metabolisers: Ref. Treatment vs Poor Metabolisers: Test Treatment; Analysis for CD 14084; Test type: Non-Inferiority or Equivalence — Equivalence range was 80% to 125%; Geometric mean ratio (%) = 104.44, 90% CI 2-sided [98.861 to 110.336], Standard Error of Mean 1.031 — Ratio calculated as poor metabolisers test treatment divided by poor metabolisers: ref. treatment

4. Secondary Outcome: Tmax of BI 409306 and Its Metabolites
Description: Time from dosing to the maximum concentration of the analyte in plasma (tmax) of BI 409306 and its metabolites CD 13896 and CD 14084
Time Frame: as for outcome 1
Population: PKS
Measure: Median (Full Range); unit: Hours
Arm/Group | Extensive Metabolisers: Ref. Treatment | Extensive Metabolisers: Test Treatment | Poor Metabolisers: Ref. Treatment | Poor Metabolisers: Test Treatment
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hours
  BI 409306 | 1.13 [0.50 to 3.00] | 1.75 [1.00 to 3.00] | 1.00 [0.50 to 4.02] | 2.00 [1.00 to 4.00]
  CD 13896 | 1.13 [0.50 to 3.00] | 2.00 [1.00 to 3.00] | 1.25 [0.50 to 4.02] | 2.00 [1.50 to 4.00]
  CD 14084 | 1.75 [1.00 to 4.00] | 2.00 [1.50 to 4.00] | 2.00 [1.00 to 4.02] | 2.50 [2.00 to 4.00]

5. Secondary Outcome: t1/2 of BI 409306 and Its Metabolites
Description: Terminal half-life of the analyte in plasma (t1/2) of BI 409306 and its metabolites CD 13896 and CD 14084
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Extensive Metabolisers: Ref. Treatment | Extensive Metabolisers: Test Treatment | Poor Metabolisers: Ref. Treatment | Poor Metabolisers: Test Treatment
Number analyzed (Participants) | 12 | 12 | 12 | 12
Hours
  BI 409306 | 1.54 (16.9) | 1.73 (27.3) | 2.87 (64.1) | 2.01 (25.2)
  CD 13896 | 2.51 (21.4) | 2.16 (21.1) | 2.26 (20.7) | 2.17 (16.8)
  CD 14084 | 3.13 (22.5) | 2.62 (10.1) | 3.21 (39.9) | 2.57 (19.7)

ADVERSE EVENTS:
Time Frame: From first trial drug intake until end of washout period or end of study visit (inclusive), up to 23 days
Description: Adverse events were analysed by the treatment being administered at the time of the adverse event.
Groups:
- Extensive Metabolizers: Itra: Participants who were extensive metabolisers receiving only 2 capsules of 100 mg itraconazole (Itra) taken orally twice daily.
- Extensive Metabolizers: BI 409306: Participants who were extensive metabolisers receiving only 1 single tablet of 25 mg BI 409306 taken orally.
- Extensive Metabolizers: Itra+BI 409306: Participants who were extensive metabolisers receiving 2 capsules of 100 mg itraconazole taken orally twice daily and 1 single tablet of 25 mg BI 409306 taken orally.
- Poor Metabolizers: Itra: Participants who were poor metabolisers receiving only 2 capsules of 100 mg itraconazole taken orally twice daily.
- Poor Metabolizers: BI 409306: Participants who were poor metabolisers receiving only 1 single tablet of 25 mg BI 409306 taken orally.
- Poor Metabolizers: Itra+BI 409306: Participants who were poor metabolisers receiving 2 capsules of 100 mg itraconazole taken orally twice daily and 1 single tablet of 25 mg BI 409306 taken orally.
Arm/Group | Extensive Metabolizers: Itra | Extensive Metabolizers: BI 409306 | Extensive Metabolizers: Itra+BI 409306 | Poor Metabolizers: Itra | Poor Metabolizers: BI 409306 | Poor Metabolizers: Itra+BI 409306
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/13 | 1/12 | 3/12 | 1/12 | 3/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extensive Metabolizers: Itra (N=13) | Extensive Metabolizers: BI 409306 (N=12) | Extensive Metabolizers: Itra+BI 409306 (N=12) | Poor Metabolizers: Itra (N=12) | Poor Metabolizers: BI 409306 (N=12) | Poor Metabolizers: Itra+BI 409306 (N=12)
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.